CLINICAL TRIAL: NCT07086742
Title: Validation of the Smart Mask V1 System and Its Measurements of SpO2 and Pulse Rate
Acronym: SMV1: PPG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pathway Medtech, LLC. (Industry)
Collaborators: Haku Technology (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: TP-SMS-0004; CIV-24-10-049534 (Other: Belgium Ministry of Health: Federal Agency for Medicines and Health Products (FAMHP))
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-06

CONDITIONS: Sleep-disordered Breathing (SDB); Sleep Apnea; Sleep Quality
Keywords: Pulse Oximeters; SpO2; Sleep apnea; postive air pressure
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The study has two Phases, both conducted using a standard 'breathe down' protocol featuring hypoxia room wherein oxygen levels are varied in 'plateaus' so that subjects' SpO2 levels are sequentially dropped from around 100% - 70% SpO2. In the first Phase, study subjects will be measured with Smart Mask, and their results (SpO2, PR) will be compared to a reference oximeter to develop a calibration for SpO2 measurements. In the second Phase, using this calibration, study subjects will be measured with Smart Mask, and their results (SpO2 only) will be compared to the CO-oximeter. For this second Phase, Smart Mask's measurements of PR will be compared to those from the reference oximeter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Non-Invasive (NI) (Experimental): The Non-Invasive (NI) study is designed to calibrate the Smart Mask's algorithms using data collected from healthy volunteers exposed to controlled, progressive hypoxia. During the study, participants lie in a supine position in a normobaric hypoxia room while breathing room air with gradually reduced oxygen levels, with the fraction of inspired oxygen (FiO2) decreasing from approximately 21% to as low as 9.5%. The Smart Mask derives SpO2 values from reflected light signals detected by its integrated sensors. Simultaneously, a benchmark pulse oximeter (Nellcor PM10N), worn on the finger, provides reference SpO2 and pulse rate (PR) values for algorithm calibration. Data from reference device are used to refine the conversion of raw photoplethysmography (PPG) signals into SpO2 and PR readings. This phase serves as a feasibility study and is a prerequisite for advancing to subsequent phase. 12 healthy subjects will be enrolled in this study.
  Interventions: Device: Smart Mask V1 System
- Invasive (IN) (Experimental): If the Non-Invasive (NI) phase demonstrates feasibility, the Invasive (IN) study will follow to validate the Smart Mask's measurements against a gold-standard method. This phase involves arterial blood gas analysis to directly measure arterial oxygen saturation (SaO2) using CO-oximetry. Participants undergo the same progressive hypoxia protocol within a controlled hypoxia room. An indwelling radial artery catheter is inserted to allow periodic arterial blood sampling at five predefined oxygen plateaus. The SaO2 values obtained from the CO-oximeter reference device (ABL90 FLEX) are then compared to the SpO2 values calculated by the Smart Mask. 24 healthy volunteers will be enrolled in this phase.
  Interventions: Device: Smart Mask V1 System

INTERVENTIONS:
Device: Smart Mask V1 System — PPG-based sensors integrated into a PAP-compatible face mask to measure SpO2 and PR.
  Other Names: Smart Mask; SMV1

SUMMARY:
The goal of this clinical study is to investigate a new medical device, the Smart Mask V1 System (herein 'Smart Mask'), and particularly its measurements of blood oxygen levels (SpO2) and pulse rate (PR) in healthy adults aged 18 to 65.

More specifically, the study is directed at answering the following questions:

* Can the Smart Mask accurately measure SpO2 levels compared to established reference devices (reference oximeters, blood gas) throughout the range of SpO2 ~ 70 - 100%?
* Can the Smart Mask accurately measure PR during the same conditions?
* Does skin pigmentation impact the accuracy of Smart Mask's measurements of SpO2 and PR.

The following reference devices will be used in the study:

* An FDA-cleared fingertip pulse oximeter (Nellcor Portable SpO2 Patient Monitoring System, PM10N)
* A laboratory-grade CO-oximeter (Radiometer ABL90 FLEX) that analyzes oxygen saturation from blood samples.

Study participants will:

* Wear the Smart Mask on their face and a fingertip pulse oximeter while lying down
* Breathe air with gradually reduced oxygen levels inside a specialized hypoxia room while being closely.
* In a second phase of the study, have a catheter inserted into a wrist artery for blood sampling to directly measure oxygen levels with the CO-oximeter.

DETAILED DESCRIPTION:
This clinical study evaluates the Smart Mask V1 System, a medical device designed to measure blood oxygen saturation (SpO2) and pulse rate (PR) using reflective photoplethysmography (PPG) sensors integrated into a face mask intended for use with positive airway pressure (PAP) therapy. The study aims to validate the accuracy of the Smart Mask's optical measurements under controlled, progressive hypoxia conditions in healthy adult volunteers.

The investigation is divided into two sequential phases; Non-Invasive (NI) and Invasive (IN) Study. All study sessions are conducted at the Complementary Medical Centre (CMC) in Genk, Belgium, within a certified normobaric hypoxia room. This room is sealed and climate-controlled, equipped with oxygen and carbon dioxide sensors to maintain a stable and safe hypoxic environment.

Hypoxia is induced gradually to reduce any discomfort or potential risk to participants. Comprehensive safety protocols are in place to protect volunteers. These include medical screening and obtaining informed consent prior to enrollment, as well as real-time monitoring by trained medical staff throughout the exposure. Immediate exit protocols are activated if a participant's SpO2 falls below 73% or if symptoms of acute mountain sickness are observed. Emergency oxygen and resuscitation equipment are readily available on-site. Additionally, participants are reminded that they may withdraw from the study at any time without penalty.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with ASA health score of I or II
* Subjects aged between ≥ 18 and ≤ 65 years.
* Subjects who have provided informed consent and are willing to comply with the study procedures.

Exclusion Criteria:

* Heavy smokers or individuals exposed to high levels of carbon monoxide resulting in elevated carboxyhemoglobin levels.
* Individuals with conditions that result in elevated methemoglobin levels.
* Individuals with hypoxia (SpO2 < 95% at 21% O2).
* Severe claustrophobia.
* Subjects known with altitude sickness.
* Subjects who are obese (BMI ≥ 35 kg/m2).
* Subjects with a known history of moderate to severe heart, lung, kidney or liver disease.
* Subjects diagnosed with moderate to severe asthma.
* Subjects with a hemoglobinopathy or history of anemia, e.g. sickle cell anemia, thalassemia, that in the investigator's opinion, would make them unsuitable for study participation.
* Subjects with any other serious systemic illness.
* Any injury, deformity, or abnormality at the sensor sites that, in the investigator's opinion, would interfere with the correct functioning of the test or reference devices.
* Subjects with a history of fainting or vasovagal response.
* Subjects with a history of sensitivity or allergy to local anesthetics or disinfectants if included in the IN study.
* Subjects diagnosed with Raynaud's disease.
* Subjects with unacceptable collateral circulation based on examination by the investigator.
* Subjects who are pregnant, lactating or trying to become pregnant.
* Subjects unable or unwilling to provide informed consent or comply with study procedures.
* Subjects with any other condition that, in the investigator's opinion, would make them unsuitable for the study.
* Subjects who refuse to remove nail polish from their index finger.
* Volunteers not willing to remove facial make-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
SpO2 Accuracy (Arms) | During each hypoxia session (90-140 minutes)
  Root mean square error (Arms) of SpO2 measured by the Smart Mask compared to SpO2 and SaO2 reference devices

CONTACTS AND LOCATIONS:
Overall Officials: Raf De Jongh, M.D., Principal Investigator — Complementair Medisch Centrum (CMC) Europe
Locations (1):
- Complementair Medisch Centrum (CMC) Europe, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No
Data collected during the study will be specifically used to develop Smart Mask, a device intended to be commercialized by the study sponsor. Thus, there does not appear to be any value or reason to share IPD.

REFERENCES:
- See also: ISO Standard document for pulse oximeters. — https://www.iso.org/standard/84775.html